CLINICAL TRIAL: NCT00947245
Title: A Randomized, Placebo-Controlled, Single and Multiple Ascending-Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of BMS-791325 in Healthy Japanese Subjects
Brief Title: Japanese Bridging Study Conducted in the United States
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: AI443-011
Record Dates: First submitted 2009-07-27; First posted 2009-07-28 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — 8-cyclohexyl-N-((dimethylamino)sulfonyl)-1,1a,2,12b-tetrahydro-11-methoxy-1a-((3-methyl-3,8-diazabicyclo(3.2.1)oct-8-yl)carbonyl)cycloprop(d)indolo(2,1-a)(2)benzazepine-5-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- BMS-791325 - Part A, Dose 1 (Experimental)
  Interventions: Drug: BMS-791325; Drug: Placebo
- BMS-791325 - Part A, Dose 2 (Experimental)
  Interventions: Drug: BMS-791325; Drug: Placebo
- BMS-791325 - Part A, Dose 3 (Experimental)
  Interventions: Drug: BMS-791325; Drug: Placebo
- BMS-791325 - Part B, Dose 1 (Experimental)
  Interventions: Drug: BMS-791325; Drug: Placebo
- BMS-791325 - Part B, Dose 2 (Experimental)
  Interventions: Drug: BMS-791325; Drug: Placebo
- BMS-791325 - Part B, Dose 3 (Experimental)
  Interventions: Drug: BMS-791325; Drug: Placebo

INTERVENTIONS:
Drug: BMS-791325 — Capsules, Oral, 300 mg, Single Dose, One day
  Arms: BMS-791325 - Part A, Dose 1
Drug: BMS-791325 — Capsules, Oral, 900 mg, Single Dose, One day
  Arms: BMS-791325 - Part A, Dose 2
Drug: BMS-791325 — Capsules, Oral, ≤1200 mg, Single Dose, One day
  Arms: BMS-791325 - Part A, Dose 3
Drug: BMS-791325 — Capsules, Oral, 300 mg, Every 12 hours, 14 days
  Arms: BMS-791325 - Part B, Dose 1
Drug: BMS-791325 — Capsules, Oral, 900 mg, once daily 14 days
  Arms: BMS-791325 - Part B, Dose 2
Drug: BMS-791325 — Capsules, Oral, ≤1200 mg, Every 12 hours or once daily, 14 days
  Arms: BMS-791325 - Part B, Dose 3
Drug: Placebo — Capsules, Oral, Single Dose, One day
  Arms: BMS-791325 - Part A, Dose 1; BMS-791325 - Part A, Dose 2; BMS-791325 - Part A, Dose 3
Drug: Placebo — Capsules, Oral, Every 12 hours, 14 days
  Arms: BMS-791325 - Part B, Dose 1
Drug: Placebo — Capsules, Oral, Once Daily, 14 days
  Arms: BMS-791325 - Part B, Dose 2
Drug: Placebo — Capsules, Oral, Every 12 hours or once daily, 14 days
  Arms: BMS-791325 - Part B, Dose 3

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics following single oral and multiple oral doses BMS-791325 in healthy Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged 20 to 49 years, with BMI of 18-30 kg/m2
* First generation Japanese. Subject born in Japan and has not lived outside of Japan for > 10 years, and subject can trace maternal and paternal Japanese ancestry

Exclusion Criteria:

* Any significant acute or chronic medical illness.
* Women who are pregnant, breastfeeding, or unwilling or unable to use an acceptable method of birth control.
* Gastrointestinal disease that may impact the absorption of study drug or that required treatment with a protocon inhibitor, antacid or H2 blocker.
* History of eczema, psoriasis, or any intermittent or active dermatitis.
* Positive for HIV or HCV

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events, physical examinations, clinical labs, ECGs, vital signs) | From time of dose to up to 14 days after last dose

SECONDARY OUTCOMES:
To measure concentration of study drug following single and multiple doses | Within 48 or 72 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Cypress, California, United States

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx